CLINICAL TRIAL: NCT03075956
Title: An Open-label, Single Center, Randomized, Two Period Study to Characterize the Safety, Tolerability and Pharmacokinetics (PK) of Estetrol (E4) After Single and Multiple Oral Doses in Healthy Female Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Estetrol (E4) After Single and Multiple Oral Doses in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MIT-Es0001-C102; 2016-001808-32 (EudraCT Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-02

CONDITIONS: Contraception; Menopause
MeSH Terms: interventions — Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5 mg E4 single-dose (Experimental): Group A: a single 5 mg E4 dose will be administered under fasted conditions during period 1.
  Interventions: Drug: 5 mg E4 single-dose
- 15 mg E4 single-dose (Experimental): Group B: a single 15 mg E4 dose will be administered under fasted conditions during period 1.
  Interventions: Drug: 15 mg E4 single-dose
- 45 mg E4 single-dose (Experimental): Group C: a single 45 mg E4 dose will be administered under fasted conditions during Period 1.
  Interventions: Drug: 45 mg E4 single-dose
- 15 mg E4 multiple-dose (Experimental): 15 mg E4 dose will be administered once daily for 14 consecutive days during Period 2.
  Interventions: Drug: 15 mg E4 multiple-dose

INTERVENTIONS:
Drug: 5 mg E4 single-dose — A single oral dose of 5 mg E4 will be administered during Period 1 of the study.
  Other Names: 5 mg estetrol
  Arms: 5 mg E4 single-dose
Drug: 15 mg E4 single-dose — A single oral dose of 15 mg E4 will be administered during Period 1 of the study.
  Other Names: 15 mg estetrol
  Arms: 15 mg E4 single-dose
Drug: 45 mg E4 single-dose — A single oral dose of 45 mg E4 will be administered once orally during Period 1 of the study
  Other Names: 45 mg estetrol
  Arms: 45 mg E4 single-dose
Drug: 15 mg E4 multiple-dose — 15 mg E4 will be administered once daily orally for 14 consecutive days during Period 2 of the study
  Other Names: 15 mg estetrol
  Arms: 15 mg E4 multiple-dose

SUMMARY:
Estetrol (E4) is being developed in two indications supporting women health care: first E4 is combined with a progestin, [drospirenone (DRSP)] and is used as a new combined oral contraceptive (COC) for the prevention of pregnancy and secondly, E4 is used alone as new hormone replacement therapy (HRT) for the treatment of menopause related symptoms.

The current clinical trial is designed to collect more detailed information about the PK profile, safety and tolerability of different dosages of E4, given orally as a solid tablet.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized, two-period, single and multiple oral dose study in 27 healthy female volunteers.

After a screening period, eligible subjects (n=27) will receive a single oral dose of 5, 15, or 45 mg E4 (Period 1). After at least 14-day washout, 18 subjects will continue the study (Period 2). They will receive 15 mg E4 once daily for 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal or premenopausal overtly healthy female subject, as determined by medical history, physical examination including breast examination, gynecological examination [including cervical smear (Pap smear)], vital signs, ECG, and laboratory tests performed.
* Between the ages of 18 and 55 years inclusive at the time of signing the informed consent.
* Between the BMI of 18 and 35 kg/m2 inclusive and body weight ≥ 45kg.
* Negative serum pregnancy test results at screening and negative urine pregnancy test results at Day -1 of Period 1.
* Venous access sufficient to allow blood sampling as per the protocol.
* Reliable and willing to be available for the duration of the study and willing to comply with the study procedures.
* Have given written informed consent (IC) approved by the relevant EC governing the site.
* Negative test results for selected drugs of abuse and cotinine at the screening visit (does not include alcohol) and at check-in for Period 1 (includes alcohol).

Exclusion Criteria:

* Use of:

  1. Any prescription drugs and/or herbal supplements acting on CYP3A4 functions, within 28 days prior to the first study dose administration until study completion.
  2. Any over-the-counter medication or dietary supplements (vitamins included) within 14 days prior to the first study dose until study completion.
* Currently breastfeeding.
* Subjects who are not in euthyroid condition.
* Known hypersensitivity to any of the investigational product ingredients.
* History of malignancy.
* History or presence of prolonged QT interval.
* Abnormal arterial tension.
* History or presence of disease of any major system organ class (e.g. cardiovascular, pulmonary, renal, hepatic, gastrointestinal, reproductive, endocrinological, neurological, psychiatric or orthopedic disease) as judged by the Investigator.
* History or presence of migraine with aura at any age or migraine without aura if > 35 years old.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
* History or presence of immunodeficiency diseases including a positive HIV test result, positive hepatitis B antigen or hepatitis C test result.
* Smokers.
* History of illicit drug or alcohol abuse within 12 months prior to first dose or evidence of such abuse.
* Donation or loss of

  * ≥ 450 mL blood within 1 month prior to initial study drug administration.
  * ≥ 250 mL blood within 2 weeks prior to initial study drug administration.
* Previous completion or withdrawal from this study.
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to study entry. Subjects who participated in an oral contraceptive clinical study, using Food and Drug Administration (FDA)/ European Union (EU) approved active ingredients, may be enrolled 2 months (60 days) after completing the preceding study.
* Sponsor, the Contract Research Organization (CRO) or Investigator's site personnel directly affiliated with this study.
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of estetrol in plasma after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
Area under the plasma concentration versus time curve from time 0 to 72 hours (AUC0-72h) of estetrol after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
Cmax at steady state (Cmaxss) of estetrol after multiple dose regimen | From Day 1 (baseline) to Day 21 of the period 2 of the study
  PK sampling on Day 1, every 2 days from Day 2 to Day 12, on Day 14, 15, 16, 17, 18, 19, 20, and 21
AUC during a dosage interval (τ) of estetrol after multiple dose regimen | From Day 1 (baseline) to Day 21 of the period 2 of the study
  PK sampling on Day 1, every 2 days from Day 2 to Day 12, on Day 14, 15, 16, 17, 18, 19, 20, and 21
Number of subjects with adverse events as a measure of safety and tolerability | From up to Day 35 before randomization to End of Study (Day 36 [+4])
  Safety will be assessed by the monitoring of adverse events (AEs), treatment emergent adverse events (TEAEs), physical examination, vital signs, electrocardiograms (ECGs), clinical laboratory test results and transvaginal ultrasound (TVUS) results

SECONDARY OUTCOMES:
AUC0-24h of estetrol after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
AUC from time 0 to infinity (AUC0-inf) of estetrol after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
Time of the maximum measured plasma concentration (Tmax) of estetrol after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
Apparent first-order terminal elimination half-life (T1/2) of estetrol after single dose regimen | From Day 1 (baseline) to Day 8 of the period 1 of the study
  PK sampling on Day 1, 2, 3, 4, 5, 6, 7 and 8
Minimum measured plasma concentration of estetrol at steady state (Cminss) after multiple dose regimen | From Day 1 (baseline) to Day 21 of the period 2 of the study
  PK sampling on Day 1, every 2 days from Day 2 to Day 12, on Day 14, 15, 16, 17, 18, 19, 20, and 21
Tmax of estetrol at steady state (Tmaxss) after multiple dose regimen | From Day 1 (baseline) to Day 21 of the period 2 of the study
  PK sampling on Day 1, every 2 days from Day 2 to Day 12, on Day 14, 15, 16, 17, 18, 19, 20, and 21

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Sviranov, Prof, Principal Investigator — Comac Medical
Locations (1):
- COMAC, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No